CLINICAL TRIAL: NCT04447755
Title: An Open-Label, Multicenter Phase 2 Basket Study to Evaluate the Antitumor Activity and Safety of Lenvatinib in Children, Adolescents, and Young Adults With Relapsed or Refractory Solid Malignancies
Brief Title: A Study of Lenvatinib (MK-7902) in Pediatric Participants With Relapsed or Refractory Solid Malignancies (MK-7902-013/E7080)
Acronym: E7080-G000-231
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7902-013; MK-7902-013 (Other: MSD); HopSkip-013 (Other: MSD); 2024-512135-80-00 (Registry Identifier: EU CT); U1111-1304-6856 (Registry Identifier: UTN); 2019-004441-33 (EudraCT Number)
Record Dates: First submitted 2020-06-23; First posted 2020-06-25 (Actual); Results first posted 2023-10-04 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Relapsed or Refractory Solid Tumors
MeSH Terms: conditions — Recurrence | interventions — lenvatinib

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Ewing Sarcoma (Experimental): Participants with Ewing sarcoma will receive lenvatinib 14 mg/m^2 once daily (QD) orally until progressive disease or unacceptable toxicity.
  Interventions: Drug: Lenvatinib
- Rhabdomyosarcoma (Experimental): Participants with rhabdomyosarcoma will receive lenvatinib 14 mg/m^2 QD orally until progressive disease or unacceptable toxicity.
  Interventions: Drug: Lenvatinib
- High Grade Glioma (Experimental): Participants with high grade glioma will receive lenvatinib 14 mg/m^2 QD orally until progressive disease or unacceptable toxicity.
  Interventions: Drug: Lenvatinib
- Diffuse Midline Glioma (Experimental): Participants with diffuse midline glioma will receive lenvatinib 14 mg/m^2 QD orally until progressive disease or unacceptable toxicity.
  Interventions: Drug: Lenvatinib
- Medulloblastoma (Experimental): Participants with medulloblastoma will receive lenvatinib 14 mg/m^2 QD orally until progressive disease or unacceptable toxicity.
  Interventions: Drug: Lenvatinib
- Ependymoma (Experimental): Participants with ependymoma will receive lenvatinib 14 mg/m^2 QD orally until progressive disease or unacceptable toxicity.
  Interventions: Drug: Lenvatinib
- Other Solid Tumors Excluding Osteosarcoma, Diffuse Midline Glioma, Medulloblastoma and Ependymoma (Experimental): Participants with other solid tumors will receive lenvatinib 14 mg/m^2 QD orally until progressive disease or unacceptable toxicity.
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib capsules administered orally at 14 mg/m^2 QD
  Other Names: MK-7902; E7080; LENVIMA

SUMMARY:
The main purpose of this study is to evaluate the antitumor activity and safety of lenvatinib (MK-7902/E7080) in children, adolescents, and young adults with relapsed or refractory solid malignancies after administration. Participants were enrolled into Ewing sarcoma (EWS), rhabdomyosarcoma (RMS), high-grade glioma (HGG), diffuse midline glioma, medulloblastoma, ependymoma, and Other Solid Tumors Excluding Osteosarcoma, diffuse midline glioma, medulloblastoma, and ependymoma cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically or cytologically documented relapsed, or refractory pediatric solid malignancy excluding osteosarcoma
* Has measurable disease as defined by Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST 1.1) or Response Assessment in Neuro-Oncology (RANO) for High Grade Glioma (HGG)
* Has a performance status defined as follows: 1) Lansky Play Score ≥50 for participants up to and including 16 years of age 2) Karnofsky performance status (KPS) ≥50 for participants >16 years of age 3) Neurologic deficits in participants with primary central nervous system (CNS) tumors must have been stable for at least 7 days prior to study enrollment
* Demonstrate adequate organ function
* No clinical evidence of nephrotic syndrome.
* Has adequate blood pressure (BP) control with or without antihypertensive medications
* Has adequate cardiac function
* Has adequate neurologic function
* Participant must have fully recovered to Common Terminology Criteria for Adverse Events, Version 5.0 (CTCAE v5.0) Grade ≤1 (except for alopecia, ototoxicity, and Grade ≤2 peripheral neuropathy) from the acute toxic effects of all prior anticancer therapy
* Male participants must agree to use approved contraception during the treatment period and for at least 7 days after the last dose of study intervention and refrain from donating sperm during this period
* Female participants are not pregnant and not breastfeeding, and are not a woman of childbearing potential (WOCBP) or are a WOCBP who agrees to follow contraceptive guidance during the treatment period and for at least 30 days after the last dose of study intervention

Exclusion Criteria:

* Has had major surgery within 3 weeks prior to Cycle 1 Day 1 (C1D1)
* Has gastrointestinal (GI) bleeding or active hemoptysis (bright red blood of at least half teaspoon) within 21 days prior to enrollment
* Has CNS tumors with a history of symptomatic tumor hemorrhage
* Has evidence of new intracranial hemorrhage of more than punctate size on MRI assessment obtained within 28 days prior to study enrollment
* Has radiographic evidence of encasement or invasion of a major blood vessel or of intratumoral cavitation
* Has evidence of untreated CNS metastases (exception: participants with primary CNS tumors and leptomeningeal disease.
* Has GI malabsorption, GI anastomosis, or any other condition that in the opinion of the investigator might affect the absorption of lenvatinib
* Has preexisting ≥Grade 3 GI or non-GI fistula
* Has any active infection requiring systemic therapy
* Known to be Human immunodeficiency virus (HIV) positive
* Known active viral hepatitis (B or C) as demonstrated by positive serology. Testing for hepatitis B or hepatitis C is required at screening only when mandated by local health authority
* Is currently participating and receiving study therapy, or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the date of allocation
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator
* Has known hypersensitivity to any component of the investigational product (lenvatinib or ingredients)
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the stud
* Has clinically significant cardiovascular disease within 6 months from first dose of study intervention, including New York Heart Association Class III or IV congestive heart failure, unstable angina, myocardial infarction, cerebral vascular accident, or cardiac arrhythmia associated with hemodynamic instability
* Has non-healing wound, tumor ulceration, unhealed or incompletely healed fracture, or a compound (open) bone fracture at the time of enrollment

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 127 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2022-09-16 (Actual); Study Completion 2025-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (49):
- United States (4):
  - Children's Hospital of Colorado ( Site 0110), Aurora, Colorado
  - Cleveland Clinic ( Site 0119), Cleveland, Ohio
  - Monroe Carell Jr. Children's Hospital at Vanderbilt ( Site 0102), Nashville, Tennessee
  - Mary Crowley Cancer Research Center ( Site 0107), Dallas, Texas
- Argentina (2):
  - Hospital Universitario Austral ( Site 0126), Pilar, Buenos Aires
  - Hospital de Niños Ricardo Gutiérrez ( Site 0125), Buenos Aires, Buenos Aires F.D.
- Australia (4):
  - Sydney Children's Hospital ( Site 0801), Randwick, New South Wales
  - Queensland Children s Hospital ( Site 0804), Brisbane, Queensland
  - Royal Childrens Hospital Melbourne ( Site 0802), Parkville, Victoria
  - Perth Children s Hospital ( Site 0803), Nedlands, Western Australia
- UZ Gent ( Site 0250), Ghent, Oost-Vlaanderen, Belgium
- Croatia (2):
  - Klinicki bolnicki centar Rijeka ( Site 0726), Rijeka, Primorje-Gorski Kotar County
  - Klinika za djecje bolesti Zagreb ( Site 0725), Zagreb, Zagreb County
- Czechia (2):
  - Fakultni Nemocnice Brno Bohunice ( Site 0651), Brno, Brno-mesto
  - Fakultni nemocnice v Motole ( Site 0650), Prague
- France (4):
  - Centre Leon-Berard ( Site 0326), Lyon, Auvergne
  - Hopital La Timone ( Site 0328), Marseille, Bouches-du-Rhone
  - Gustave Roussy ( Site 0327), Villejuif, Val-de-Marne
  - Institut Curie ( Site 0325), Paris
- Guatemala (2):
  - Unidad Nacional de Oncologia Pediatrica ( Site 0176), Guatemala City
  - Medi-K Cayala ( Site 0177), Guatemala City
- Hungary (3):
  - Borsod-Abauj-Zemplen Megyei Korhaz es Egyetemi OktatoKorhaz ( Site 0678), Miskolc, Borsod-Abauj Zemplen county
  - Semmelweis University ( Site 0675), Budapest
  - Debreceni Egyetem Klinikai Kozpont ( Site 0677), Debrecen
- Chaim Sheba Medical Center ( Site 0500), Ramat Gan, Israel
- Italy (5):
  - IRCCS Ospedale Pediatrico Bambino Gesu ( Site 0410), Rome, Roma
  - A.O.Universitaria Meyer-Oncology & Haematology Unit ( Site 0400), Florence, Tuscany
  - Istituto Giannina Gaslini ( Site 0411), Genova
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano ( Site 0401), Milan
  - Ospedale Infantile Regina Margherita ( Site 0412), Torino
- Starship Childrens Hospital ( Site 0826), Auckland, New Zealand
- Clinica Anglo Americana ( Site 0203), San Isidro, Lima region, Peru
- Russia (3):
  - Dmitry Rogachev National Research Center ( Site 0550), Moscow, Moscow
  - St.Petersburg State Medical Univ. n.a. acad. I.P.Pavlov ( Site 0554), Saint Petersburg, Sankt-Peterburg
  - Clinical Research Center of specialized types medical care-Oncology ( Site 0553), Saint Petersburg, Sankt-Peterburg
- Serbia (2):
  - Institute for Oncology and Radiology of Serbia ( Site 0780), Belgrade, Beograd
  - Univerzitetska decja klinika ( Site 0782), Belgrade, Beograd
- South Africa (3):
  - Wits Clinical Research ( Site 0579), Soweto, Gauteng
  - Cancercare Rondebosch Oncology ( Site 0575), Cape Town, Western Cape
  - Tygerberg Hospital ( Site 0578), Parow, Western Cape
- South Korea (2):
  - Asan Medical Center ( Site 0876), Songpagu, Seoul
  - Seoul National University Hospital ( Site 0875), Seoul
- Spain (2):
  - Hospital Universitario Sant Joan de Deu ( Site 0476), Esplugues de Llobregat, Barcelona
  - Hospital Nino Jesus ( Site 0477), Madrid
- Skanes Universitetssjukhus Lund. ( Site 0525), Lund, Skåne County, Sweden
- Turkey (Türkiye) (4):
  - Hacettepe Universitesi Tip Fakultesi ( Site 0603), Ankara
  - Istanbul Universitesi Onkoloji Enstitusu ( Site 0600), Istanbul
  - Ege Universitesi Tip Fakultesi ( Site 0601), Izmir
  - Dokuz Eylul Universitesi Arastirma Uygulama Hastanesi ( Site 0602), Izmir

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] Gaspar N, Campbell-Hewson Q, Gallego Melcon S, Locatelli F, Venkatramani R, Hecker-Nolting S, Gambart M, Bautista F, Thebaud E, Aerts I, Morland B, Rossig C, Canete Nieto A, Longhi A, Lervat C, Entz-Werle N, Strauss SJ, Marec-Berard P, Okpara CE, He C, Dutta L, Casanova M. Phase I/II study of single-agent lenvatinib in children and adolescents with refractory or relapsed solid malignancies and young adults with osteosarcoma (ITCC-050)☆. ESMO Open. 2021 Oct;6(5):100250. doi: 10.1016/j.esmoop.2021.100250. Epub 2021 Sep 22. PMID 34562750
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26352&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited to tumor cohorts of Ewing Sarcoma, Rhabdomyosarcoma, High Grade Glioma, and Other Solid Tumors Excluding Osteosarcoma. Enrollment to the protocol pre-specified tumor cohort of "Other Solid Tumors Excluding Osteosarcoma" was further expanded into categories of Diffuse midline glioma, Medulloblastoma, and Ependymoma.
Groups:
- Ewing Sarcoma: Participants with Ewing sarcoma received lenvatinib 14 mg/m^2 once daily (QD) orally until progressive disease or unacceptable toxicity.
- Rhabdomyosarcoma: Participants with rhabdomyosarcoma received lenvatinib 14 mg/m^2 QD orally until progressive disease or unacceptable toxicity.
- High Grade Glioma: Participants with high grade glioma received lenvatinib 14 mg/m^2 QD orally until progressive disease or unacceptable toxicity.
- Diffuse Midline Glioma: Participants with diffuse midline glioma received lenvatinib 14 mg/m^2 QD orally until progressive disease or unacceptable toxicity.
- Medulloblastoma: Participants with medulloblastoma received lenvatinib 14 mg/m^2 QD orally until progressive disease or unacceptable toxicity.
- Ependymoma: Participants with ependymoma received lenvatinib 14 mg/m^2 QD orally until progressive disease or unacceptable toxicity.
- Other Solid Tumors Excluding Osteosarcoma, Diffuse Midline Glioma, Medulloblastoma and Ependymoma: Participants with other solid tumors received lenvatinib 14 mg/m^2 QD orally until progressive disease or unacceptable toxicity.
Period: Overall Study
Arm/Group | Ewing Sarcoma | Rhabdomyosarcoma | High Grade Glioma | Diffuse Midline Glioma | Medulloblastoma | Ependymoma | Other Solid Tumors Excluding Osteosarcoma, Diffuse Midline Glioma, Medulloblastoma and Ependymoma
Started | 9 | 17 | 8 | 9 | 9 | 9 | 66
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 9 | 17 | 8 | 9 | 9 | 9 | 66
Not completed — Death | 9 | 16 | 8 | 9 | 8 | 9 | 55
Not completed — Withdrawal by Parent/Guardian | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 1 | 0 | 10
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ewing Sarcoma | Rhabdomyosarcoma | High Grade Glioma | Diffuse Midline Glioma | Medulloblastoma | Ependymoma | Other Solid Tumors Excluding Osteosarcoma, Diffuse Midline Glioma, Medulloblastoma and Ependymoma | Total
Number analyzed (Participants) | 9 | 17 | 8 | 9 | 9 | 9 | 66 | 127
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.8 (4.0) | 13.1 (4.7) | 14.0 (3.1) | 10.0 (5.2) | 13.2 (4.5) | 8.7 (5.7) | 13.1 (5.6) | 12.7 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 4 | 8 | 3 | 4 | 32 | 60
  Male | 7 | 10 | 4 | 1 | 6 | 5 | 34 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 0 | 1 | 0 | 9 | 13
  Not Hispanic or Latino | 5 | 11 | 6 | 4 | 2 | 6 | 43 | 77
  Unknown or Not Reported | 3 | 4 | 2 | 5 | 6 | 3 | 14 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 3
  Asian | 3 | 2 | 1 | 3 | 0 | 0 | 13 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4
  White | 3 | 10 | 4 | 2 | 2 | 7 | 35 | 63
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 2 | 4 | 3 | 4 | 6 | 2 | 11 | 32

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) At Week 16 Per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1) or Response Assessment in Neuro-Oncology (RANO) Criteria (for High Grade Glioma [HGG] Only), by Investigator Assessment
Description: ORR at Week 16 was defined as the percentage of participants with a confirmed complete response (CR: disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters [SOD] of target lesions, taking as reference the baseline SOD) as assessed by the investigator per RECIST 1.1 at 16 Weeks. For participants with HGG, response was assessed according to RANO criteria whereby overall response is based on both radiographic response (CR: disappearance of all target lesions, PR: sum of products of diameters [SPD] decreased by ≥ 50% from baseline value) and clinical performance status with steroid dose information.
Time Frame: Up to 16 weeks
Population: All participants who had measurable disease present at baseline and at least one efficacy assessment, unless they discontinued prior to the first efficacy assessment due to progressive disease.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ewing Sarcoma | Rhabdomyosarcoma | High Grade Glioma | Diffuse Midline Glioma | Medulloblastoma | Ependymoma | Other Solid Tumors Excluding Osteosarcoma, Diffuse Midline Glioma, Medulloblastoma and Ependymoma
Number analyzed (Participants) | 9 | 17 | 6 | 9 | 9 | 9 | 65
Percentage of Participants | 22.2 [2.8 to 60.0] | 11.8 [1.5 to 36.4] | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 33.6] | 7.7 [2.5 to 17.0]

2. Secondary Outcome: ORR Per RECIST 1.1 or RANO Criteria (for HGG Only), by Investigator Assessment
Description: ORR was defined as the percentage of participants with a confirmed complete response (CR: disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD) as assessed by the investigator per RECIST 1.1. For participants with HGG, response was assessed according to RANO criteria whereby overall RANO response is based on both radiographic response (CR: disappearance of all target lesions, PR: SPD decreased by ≥ 50% from baseline value) and clinical performance status with steroid dose information.
Time Frame: Up to approximately 21 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ewing Sarcoma | Rhabdomyosarcoma | High Grade Glioma | Diffuse Midline Glioma | Medulloblastoma | Ependymoma | Other Solid Tumors Excluding Osteosarcoma, Diffuse Midline Glioma, Medulloblastoma and Ependymoma
Number analyzed (Participants) | 9 | 17 | 6 | 9 | 9 | 9 | 65
Percentage of Participants | 22.2 [2.8 to 60.0] | 11.8 [1.5 to 36.4] | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 33.6] | 7.7 [2.5 to 17.0]

3. Secondary Outcome: Progression Free Survival (PFS) Per RECIST 1.1 or RANO (for HGG Only), by Investigator Assessment
Description: PFS was defined as the time from the date of the first administration of study drug until the date of first documentation of progressive disease (PD) per RECIST 1.1 or RANO (for HGG) or death (whichever occurs first).
Time Frame: Up to approximately 21 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ewing Sarcoma | Rhabdomyosarcoma | High Grade Glioma | Diffuse Midline Glioma | Medulloblastoma | Ependymoma | Other Solid Tumors Excluding Osteosarcoma, Diffuse Midline Glioma, Medulloblastoma and Ependymoma
Number analyzed (Participants) | 9 | 17 | 6 | 9 | 9 | 9 | 65
Months | 3.0 [0.3 to 9.3] | 2.6 [1.2 to 5.6] | 1.9 [1.4 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | 1.8 [0.5 to 4.9] | 3.4 [0.5 to 8.5] | 2.5 [1.2 to 7.4] | 3.8 [3.2 to 5.7]

4. Secondary Outcome: Best Overall Response (BOR) Per RECIST 1.1 or RANO (for HGG Only), by Investigator Assessment
Description: BOR is defined as the participant's best confirmed response (CR or PR) over the treatment period as assessed by the investigator per RECIST 1.1 or RANO. As per RECIST 1.1, CR is defined as disappearance of all target lesions and PR is defined as at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD. For participants with HGG, response will be assessed according to RANO criteria whereby overall RANO response is based on both radiographic response (CR: disappearance of all target lesions, PR: SPD decreased by ≥ 50% from baseline value) and clinical performance status with steroid dose information.
Time Frame: Up to approximately 21 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ewing Sarcoma | Rhabdomyosarcoma | High Grade Glioma | Diffuse Midline Glioma | Medulloblastoma | Ependymoma | Other Solid Tumors Excluding Osteosarcoma, Diffuse Midline Glioma, Medulloblastoma and Ependymoma
Number analyzed (Participants) | 9 | 17 | 6 | 9 | 9 | 9 | 65
Percentage of Participants | 22.2 [2.8 to 60.0] | 11.8 [1.5 to 36.4] | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 33.6] | 7.7 [2.5 to 17.0]

5. Secondary Outcome: Duration of Response (DOR) Per RECIST 1.1 or RANO (for HGG Only), by Investigator Assessment
Description: DOR was defined as the time from the date of the first documented CR or PR to the date first documentation of progressive disease or death (whichever occurs first). As per RECIST 1.1, CR was defined as disappearance of all target lesions and PR was defined as at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD. For participants with HGG, response will be assessed according to RANO criteria whereby overall RANO response is based on both radiographic response (CR: disappearance of all target lesions, PR: SPD decreased by ≥ 50% from baseline value) and clinical performance status with steroid dose information.
Time Frame: Up to approximately 21 months
Population: All participants who had measurable disease present at baseline and at least one efficacy assessment, unless they discontinued prior to the first efficacy assessment due to progressive disease, and demonstrated CR or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ewing Sarcoma | Rhabdomyosarcoma | High Grade Glioma | Diffuse Midline Glioma | Medulloblastoma | Ependymoma | Other Solid Tumors Excluding Osteosarcoma, Diffuse Midline Glioma, Medulloblastoma and Ependymoma
Number analyzed (Participants) | 2 | 2 | 0 | 0 | 0 | 0 | 5
Months | NA [5.7 to NA] — NA = Median and upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse. | 4.6 [3.7 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse. |  |  |  |  | 4.6 [3.7 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse.

6. Secondary Outcome: Disease Control Rate (DCR) Per RECIST 1.1 or RANO (for HGG Only), by Investigator Assessment
Description: DCR was defined as a BOR of CR or PR, or stable disease (SD). To be assigned a BOR of SD, the time from the first administration of study drug until the date of documented SD should be ≥7 weeks. As per RECIST 1.1, CR was defined as disappearance of all target lesions, PR was defined as at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD, and SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. For participants with HGG, response was assessed according to RANO criteria whereby overall response was based on both radiographic response (CR: disappearance of all target lesions, PR: SPD decreased by ≥ 50% from baseline value and SD: SPD <50% decreased from baseline, but <25% increased from nadir) and clinical performance status with steroid dose information.
Time Frame: Up to approximately 21 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ewing Sarcoma | Rhabdomyosarcoma | High Grade Glioma | Diffuse Midline Glioma | Medulloblastoma | Ependymoma | Other Solid Tumors Excluding Osteosarcoma, Diffuse Midline Glioma, Medulloblastoma and Ependymoma
Number analyzed (Participants) | 9 | 17 | 6 | 9 | 9 | 9 | 65
Percentage of Participants | 66.7 [29.9 to 92.5] | 52.9 [27.8 to 77.0] | 33.3 [4.3 to 77.7] | 22.2 [2.8 to 60.0] | 55.6 [21.2 to 86.3] | 55.6 [21.2 to 86.3] | 64.6 [51.8 to 76.1]

7. Secondary Outcome: Clinical Benefit Rate (CBR) Per RECIST 1.1 or RANO (for HGG Only), by Investigator Assessment
Description: CBR was defined as a BOR of CR or PR, or durable SD (Duration of SD should be ≥23 weeks since the first dose of the study treatment. As per RECIST 1.1, CR was defined as disappearance of all target lesions, PR was defined as at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD and SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. For participants with HGG, response is assessed according to RANO criteria whereby overall response was based on both radiographic response (CR: disappearance of all target lesions, PR: SPD decreased by ≥ 50% from baseline value and SD: SPD <50% decreased from baseline, but <25% increased from nadir) and clinical performance status with steroid dose information.
Time Frame: Up to approximately 21 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ewing Sarcoma | Rhabdomyosarcoma | High Grade Glioma | Diffuse Midline Glioma | Medulloblastoma | Ependymoma | Other Solid Tumors Excluding Osteosarcoma, Diffuse Midline Glioma, Medulloblastoma and Ependymoma
Number analyzed (Participants) | 9 | 17 | 6 | 9 | 9 | 9 | 65
Percentage of Participants | 33.3 [7.5 to 70.1] | 29.4 [10.3 to 56.0] | 0.0 [0.0 to 45.9] | 11.1 [0.3 to 48.2] | 44.4 [13.7 to 78.8] | 33.3 [7.5 to 70.1] | 40.0 [28.0 to 52.9]

8. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experienced at least one AE is reported.
Time Frame: Up to approximately 50 months
Population: All participants who received at least one dose of study treatment were analyzed.
Measure: Number; unit: Participants
Arm/Group | Ewing Sarcoma | Rhabdomyosarcoma | High Grade Glioma | Diffuse Midline Glioma | Medulloblastoma | Ependymoma | Other Solid Tumors Excluding Osteosarcoma, Diffuse Midline Glioma, Medulloblastoma and Ependymoma
Number analyzed (Participants) | 9 | 17 | 8 | 9 | 9 | 9 | 66
Participants | 9 | 17 | 8 | 9 | 9 | 8 | 66

9. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinued study treatment due to an AE is reported.
Time Frame: Up to approximately 38 months
Population: All participants who received at least one dose of study treatment were analyzed.
Measure: Number; unit: Participants
Arm/Group | Ewing Sarcoma | Rhabdomyosarcoma | High Grade Glioma | Diffuse Midline Glioma | Medulloblastoma | Ependymoma | Other Solid Tumors Excluding Osteosarcoma, Diffuse Midline Glioma, Medulloblastoma and Ependymoma
Number analyzed (Participants) | 9 | 17 | 8 | 9 | 9 | 9 | 66
Participants | 1 | 0 | 0 | 0 | 1 | 2 | 6

10. Secondary Outcome: Palatability Questionnaire For Lenvatinib Suspension Formulation: Participant Responses by Taste Category
Description: A hedonic Visual Analog Scale (VAS) was used to assess taste likability or "palatability" of a lenvatinib suspension formulated with water or apple juice. Participants scored each category on a scale from 1-7 ranging from super bad (score = 1) to super good (score = 7). As pre-specified by the supplemental Statistical Analysis Plan (sSAP), all participants who received suspension formulation were evaluated for palatability and acceptability of the suspension formulation, and data were summarized in an overall safety analysis set irrespective of tumor type. The palatability score based on the taste category is presented.
Time Frame: Cycle 1 Day 1 (cycle = 28 days)
Population: Per protocol, all participants who received suspension formulation were analyzed. Data were summarized in an overall safety analysis set irrespective of tumor type.
Measure: Number; unit: Participants
Groups:
- All Tumor Types: Participants received lenvatinib 14 mg/m^2 once daily (QD) orally until progressive disease or unacceptable toxicity.
Arm/Group | All Tumor Types
Number analyzed (Participants) | 10
Participants
  Super Bad | 1
  Really Bad | 0
  Bad | 2
  Maybe Good or Maybe Bad | 5
  Good | 1
  Really Good | 0
  Super Good | 1

11. Secondary Outcome: Palatability Questionnaire For Lenvatinib Suspension Formulation: Participant Responses by Appearance Category
Description: A hedonic VAS was used to assess taste likability or "palatability" of a lenvatinib suspension formulated with water or apple juice. Participants scored each category on a scale from 1-7 ranging from super bad (score = 1) to super good (score = 7). As pre-specified by the sSAP, all participants who received suspension formulation were evaluated for palatability and acceptability of the suspension formulation, and data were summarized in an overall safety analysis set irrespective of tumor type. The palatability score based on the appearance category is presented.
Time Frame: Cycle 1 Day 1 (cycle = 28 days)
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | All Tumor Types
Number analyzed (Participants) | 10
Participants
  Super Bad | 0
  Really Bad | 0
  Bad | 1
  Maybe Good or Maybe Bad | 5
  Good | 2
  Really Good | 0
  Super Good | 2

12. Secondary Outcome: Palatability Questionnaire For Lenvatinib Suspension Formulation: Participant Responses by Smell Category
Description: A hedonic VAS was used to assess taste likability or "palatability" of a lenvatinib suspension formulated with water or apple juice. Participants scored each category on a scale from 1-7 ranging from super bad (score = 1) to super good (score = 7). As pre-specified by the sSAP, all participants who received suspension formulation were evaluated for palatability and acceptability of the suspension formulation, and data were summarized in an overall safety analysis set irrespective of tumor type. The palatability score based on the smell category is presented.
Time Frame: Cycle 1 Day 1 (cycle = 28 days)
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | All Tumor Types
Number analyzed (Participants) | 10
Participants
  Super Bad | 0
  Really Bad | 0
  Bad | 0
  Maybe Good or Maybe Bad | 8
  Good | 1
  Really Good | 0
  Super Good | 1

13. Secondary Outcome: Palatability Questionnaire For Lenvatinib Suspension Formulation: Participant Responses by Mouth Feel Category
Description: A hedonic VAS was used to assess taste likability or "palatability" of a lenvatinib suspension formulated with water or apple juice. Participants scored each category on a scale from 1-7 ranging from super bad (score = 1) to super good (score = 7). As pre-specified by the sSAP, all participants who received suspension formulation were evaluated for palatability and acceptability of the suspension formulation, and data were summarized in an overall safety analysis set irrespective of tumor type. The palatability score based on the mouth feel category is presented.
Time Frame: Cycle 1 Day 1 (cycle = 28 days)
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | All Tumor Types
Number analyzed (Participants) | 10
Participants
  Super Bad | 0
  Really Bad | 1
  Bad | 2
  Maybe Good or Maybe Bad | 4
  Good | 1
  Really Good | 2
  Super Good | 0

14. Secondary Outcome: Palatability Questionnaire For Lenvatinib Suspension Formulation: Participant Responses by Overall Acceptability Category
Description: A hedonic VAS was used to assess taste likability or "palatability" of a lenvatinib suspension formulated with water or apple juice. Participants scored each category on a scale from 1-7 ranging from super bad (score = 1) to super good (score = 7). As pre-specified by the sSAP, all participants who received suspension formulation were evaluated for palatability and acceptability of the suspension formulation, and data were summarized in an overall safety analysis set irrespective of tumor type. The palatability score based on the overall acceptability category is presented.
Time Frame: Cycle 1 Day 1 (cycle = 28 days)
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | All Tumor Types
Number analyzed (Participants) | 10
Participants
  Super Bad | 0
  Really Bad | 1
  Bad | 1
  Maybe Good or Maybe Bad | 3
  Good | 3
  Really Good | 1
  Super Good | 1

15. Secondary Outcome: Area Under the Concentration-Time Curve of Lenvatinib at Steady State (AUCss)
Description: Blood samples were taken predose and at specified times postdose on Days 1-28 to determine the AUCss of Lenvatinib.
Time Frame: Cycle 1 Day 1 (0.5-4 and 6-10 hours post-dose), Cycle 1 Day 15 (pre-dose, 0.5-4, and 6-10 hours post-dose), and Cycle 2 Day 1 (pre-dose and 2-12 hours post-dose). A cycle is 28 days.
Population: All participants who received at least one dose of study treatment and had at least one measurable postdose plasma concentration with an adequately documented dosing history were analyzed. Lenvatinib exposures are reported by the four protocol pre-specified cohorts at the time of enrollment (EWS, RMS, HGG, and Other Solid Tumors excluding Osteosarcoma). For the purposes of the analysis, AUCss was reported for participants with "Other Solid Tumors" irrespective of tumor type.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/ml
Groups:
- Other Solid Tumors Excluding Osteosarcoma: Participants with other solid tumors received lenvatinib 14 mg/m^2 QD orally until progressive disease or unacceptable toxicity.
Arm/Group | Ewing Sarcoma | Rhabdomyosarcoma | High Grade Glioma | Other Solid Tumors Excluding Osteosarcoma
Number analyzed (Participants) | 9 | 17 | 8 | 91
ng*hr/ml | 5896 (31.2) | 3915 (32.9) | 3660 (43.5) | 4990 (53.2)

ADVERSE EVENTS:
Time Frame: Up to approximately 50 months
Description: The analysis population for All-Cause Mortality included all allocated participants. The safety analysis population included all allocated participants who received at least one dose of study treatment. Per protocol, disease progression of cancer under study was not considered an AE unless considered related to study treatment. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" & "Disease progression" not related to study treatment are excluded as AEs.
Arm/Group | Ewing Sarcoma | Rhabdomyosarcoma | High Grade Glioma | Diffuse Midline Glioma | Medulloblastoma | Ependymoma | Other Solid Tumors Excluding Osteosarcoma, Diffuse Midline Glioma, Medulloblastoma and Ependymoma
All-Cause Mortality (participants affected / at risk) | 9/9 | 17/17 | 8/8 | 9/9 | 8/9 | 9/9 | 55/66
Serious Adverse Events (participants affected / at risk) | 4/9 | 5/17 | 6/8 | 4/9 | 4/9 | 4/9 | 39/66
Other Adverse Events (participants affected / at risk) | 9/9 | 17/17 | 6/8 | 9/9 | 9/9 | 7/9 | 66/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ewing Sarcoma (N=9) | Rhabdomyosarcoma (N=17) | High Grade Glioma (N=8) | Diffuse Midline Glioma (N=9) | Medulloblastoma (N=9) | Ependymoma (N=9) | Other Solid Tumors Excluding Osteosarcoma, Diffuse Midline Glioma, Medulloblastoma and Ependymoma (N=66)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orbital compartment syndrome (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Complication associated with device (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device related sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (5)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Neurogenic bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngeal fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (11)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ewing Sarcoma (N=9) | Rhabdomyosarcoma (N=17) | High Grade Glioma (N=8) | Diffuse Midline Glioma (N=9) | Medulloblastoma (N=9) | Ependymoma (N=9) | Other Solid Tumors Excluding Osteosarcoma, Diffuse Midline Glioma, Medulloblastoma and Ependymoma (N=66)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 13 (15)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (13)
Cardiac dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (5)
Ear haemorrhage (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Excessive cerumen production (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 7 (8) | 8 (8) | 4 (4) | 7 (7) | 7 (7) | 5 (5) | 45 (47)
Corneal erosion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Eyelid ptosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lagophthalmos (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Strabismus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (4) | 6 (9) | 1 (1) | 0 (0) | 2 (5) | 1 (3) | 14 (18)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 4 (5) | 2 (3) | 2 (2) | 3 (3) | 0 (0) | 11 (12)
Diarrhoea (Gastrointestinal disorders) | 5 (13) | 6 (7) | 0 (0) | 0 (0) | 4 (8) | 3 (7) | 22 (41)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (10)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 3 (4) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 13 (13)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 4 (4)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (8) | 7 (7) | 1 (1) | 2 (2) | 4 (5) | 2 (2) | 18 (27)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 3 (3)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chest pain (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 5 (5) | 0 (0) | 13 (14)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 9 (12)
Xerosis (General disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cytolysis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asymptomatic bacteriuria (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (7)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lip infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (5)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pyuria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 1 (3) | 0 (0) | 7 (8)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Medication error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urethral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (9) | 3 (3) | 1 (1) | 0 (0) | 3 (5) | 1 (1) | 15 (22)
Amylase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (7)
Aspartate aminotransferase increased (Investigations) | 3 (6) | 5 (5) | 2 (2) | 0 (0) | 2 (4) | 2 (2) | 13 (15)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (7)
Blood bilirubin increased (Investigations) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 4 (5)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 6 (7)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Blood urea increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram T wave abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 3 (4)
Haemoglobin increased (Investigations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 3 (5)
Platelet count decreased (Investigations) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 4 (5) | 1 (1) | 14 (16)
Protein total decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroxine free increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 19 (19)
White blood cell count decreased (Investigations) | 1 (3) | 1 (1) | 1 (1) | 0 (0) | 2 (6) | 0 (0) | 6 (7)
Decreased appetite (Metabolism and nutrition disorders) | 5 (6) | 7 (7) | 2 (2) | 3 (3) | 3 (3) | 1 (1) | 18 (22)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (9)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 8 (10)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4) | 1 (1) | 1 (1) | 3 (4) | 1 (1) | 7 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (7) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 5 (7)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 9 (13)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour exudation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Coma (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diplegia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 4 (6) | 0 (0) | 1 (1) | 3 (3) | 3 (5) | 9 (9)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemiplegia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyporeflexia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotonia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasticity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myoclonus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neurological decompensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petit mal epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Quadriparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bradyphrenia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Poor quality sleep (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glycosuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Proteinuria (Renal and urinary disorders) | 2 (2) | 5 (6) | 0 (0) | 3 (3) | 2 (3) | 1 (2) | 28 (38)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast induration (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (6)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 9 (10)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 4 (4)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 6 (6)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (7)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 7 (9)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 3 (4) | 6 (7) | 2 (3) | 5 (5) | 3 (3) | 3 (3) | 27 (33)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-08): https://cdn.clinicaltrials.gov/large-docs/55/NCT04447755/Prot_SAP_000.pdf